CLINICAL TRIAL: NCT02695862
Title: To Assess Safety and Efficacy of Bolus Versus Continuous Infusion of Terlipressin in Acute Variceal Bleeding: A Randomized Comparison
Brief Title: To Assess Safety and Efficacy of Bolus Versus Continuous Infusion of Terlipressin in Acute Variceal Bleeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-AVB-001
Record Dates: First submitted 2016-02-25; First posted 2016-03-01 (Estimated); Last update posted 2019-09-04 (Actual); Status verified 2017-09

CONDITIONS: Acute Variceal Bleeding
MeSH Terms: interventions — Terlipressin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bolus Terlipressin (Experimental): Injection terlipressin after 2 mg bolus it will be given 2 mg QID
  Interventions: Drug: Terlipressin
- Terlipressin continuous(4mg/24hours) (Active Comparator): Injection terlipressin after 2 mg bolus it will be given 4 mg over 24 hours,and dose will be titrated as per HVPG (Hepatic Venous Pressure Gradient)
  Interventions: Drug: Terlipressin

INTERVENTIONS:
Drug: Terlipressin

SUMMARY:
The study is single centered; prospective, parallel arm randomized controlled trial.The patients will be who presented to Institute of Liver & Biliary Sciences with esophageal variceal bleeding or develop esophageal bleeding during hospital stay. All patients will be managed with continuous non-invasive cardiac and hemodynamic monitoring including cardiac rhythm, pulse rate, blood pressure, and oxygen saturation. Hemoglobin (Hb) will checked every 6 h for the initial 48 h and then every 12 h till discharge. Likewise, serum creatinine will checked daily. Packed red blood cells will be transfused to maintain target Hb of ⩾8 g/dl. Patients will be started on IV Proton Pump Inhibitor, with bolus dose of terlipressin (2mg) followed by Endoscopic variceal ligation. All patients will received prophylactic antibiotics; antibiotics will be stopped if there will no other indication to continue. After confirmation of EVB (Esophageal Variceal Bleeding) and successful initial hemostasis with emergency EVBL (Endoscopic Variceal Band ligation), patients will be randomly assigned into Group -A (Bolus terlipressin at 2mg every 4hourly) and Group-B (Continuous infusion of terlipressin @ 4mg/24hour initially) therapy for esophageal varices . They will then undergo HVPG (Hepatic Venous Pressure Gradient) measurement at baseline, 12hours and 24hours. Patient in continuous group will titrate dose. accordingly to HVPG (Hepatic Venous Pressure Gradient) measurement at 12 and 24 hours. At 24 hours patient will be directed to receive either TIPS (Transjugular Intrahepatic Portosystemic Shunt) or will continue Terlipressin for 48 hours.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with only acute esophageal variceal bleeding (as defined by Asian pacific Association for the study of Liver Disease)
* Informed consent to participate in the study
* Age 18 to 70 years

Exclusion Criteria:

* Pregnant and lactation
* Prior treatment with any vasoactive drugs
* Significant heart or respiratory failure
* Peripheral arteriopathy clinically significant
* Previous heart stroke or significant alteration of the Electrocardiogram
* Hemodynamically unstable
* Refusal to participate in the study
* Hypertension

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2016-05-05 (Actual); Primary Completion 2017-12-10 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Reduction of HVPG (hepatic venous pressure gradient) at 24 hours >10% | 24 hours

SECONDARY OUTCOMES:
Death in both groups | 42 days
Terlipressin related complications in both groups | 72 hours
Rebleed within 42 days | 42 days
number of blood transfusion requirement at 5 days | 5 days
Incidence of ischaemic hepatitis within 5 days | 5 days
Incidence of post bleed acute kidney injury within 5 days | 5 days
Incidence of post EVL(endoscopic band ligation) ulcer bleed within 5 days | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Dr Shakti P Choudhury, MD, Principal Investigator — Institute of Liver and Biliary Sciences
Locations (1):
- Institute of liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Arora V, Choudhary SP, Maiwall R, Vijayaraghavan R, Jindal A, Kumar G, Sarin SK. Low-dose continuous terlipressin infusion is effective and safer than intravenous bolus injections in reducing portal pressure and control of acute variceal bleeding. Hepatol Int. 2023 Feb;17(1):131-138. doi: 10.1007/s12072-022-10416-6. Epub 2022 Dec 21. PMID 36542261